CLINICAL TRIAL: NCT05160558
Title: A Phase 1, Blinded, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of BIIB132 Administered Intrathecally to Adults With Spinocerebellar Ataxia 3
Brief Title: A Pharmacokinetics and Safety Study of BIIB132 in Adults With Spinocerebellar Ataxia 3
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 260SA101; 2021-002223-37 (EudraCT Number)
Record Dates: First submitted 2021-12-07; First posted 2021-12-16 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Spinocerebellar Ataxia Type 3
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: BIIB132 Dose 1 or Matching Placebo (Experimental): Participants will be randomized to receive BIIB132 Dose 1 or matching placebo, intrathecally (IT), every 4 weeks (Q4W), up to Day 85.
  Interventions: Drug: BIIB132; Drug: BIIB132-Matching Placebo
- Cohort 2: BIIB132 Dose 2 or Matching Placebo (Experimental): Participants will be randomized to receive BIIB132 Dose 2 or matching placebo, IT, Q4W, up to Day 85.
  Interventions: Drug: BIIB132; Drug: BIIB132-Matching Placebo
- Cohort 3: BIIB132 Dose 3 or Matching Placebo (Experimental): Participants will be randomized to receive BIIB132 Dose 3 or matching placebo, IT, Q4W, up to Day 85.
  Interventions: Drug: BIIB132; Drug: BIIB132-Matching Placebo
- Cohort 4: BIIB132 Dose 4 or Matching Placebo (Experimental): Participants will be randomized to receive BIIB132 Dose 4 or matching placebo, IT, Q4W, up to Day 85.
  Interventions: Drug: BIIB132; Drug: BIIB132-Matching Placebo
- Cohort 5: BIIB132 Dose 5 or Matching Placebo (Experimental): Participants will be randomized to receive BIIB132 Dose 5 or matching placebo, IT, either Q4W or every 12 weeks (Q12W), up to Day 85 or every 8 weeks (Q8W) up to Day 57.
  Interventions: Drug: BIIB132; Drug: BIIB132-Matching Placebo

INTERVENTIONS:
Drug: BIIB132 — Administered as specified in the treatment arm
Drug: BIIB132-Matching Placebo — Administered as specified in the treatment arm

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple ascending doses of BIIB132 administered via intrathecal (IT) injection to participants with spinocerebellar ataxia type 3 (SCA3). The secondary objective of this study is to characterize the multiple-dose pharmacokinetics (PK) of BIIB132 administered via IT injection to participants with SCA3.

DETAILED DESCRIPTION:
BIIB132 is an investigational anti-sense oligonucleotide developed to target ataxin-3 (ATXN3) pre-messenger ribonucleic acid (pre-mRNA). Preclinical studies have shown that lowering of ATXN3 protein is associated with decreased progression of SCA3-like disease. This trial consists of a blinded 12 week study period with a 26 week follow up period to evaluate the safety and tolerability of intrathecal BIIB132 and to assess the effect on treatment response biomarkers in symptomatic SCA3 participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of SCA3 with CAG repeats ≥60 in ATXN3 gene.
* Symptomatic ataxia with a screening Scale for Assessment and Rating of Ataxia (SARA) score 3 to 15 (still ambulatory) and a minimum SARA gait subscore of 1.
* Able to ambulate 8 m independently without any assistive device.
* Treatment naïve or on a stable dose of symptomatic therapy for a minimum of 4 weeks prior to screening.

Key Exclusion Criteria:

* Unstable psychiatric illness or untreated major depression within 90 days before screening.
* History or screening magnetic resonance imaging (MRI) results show evidence of structural abnormalities that could contribute to the participant's clinical state other than findings typical of SCA3 or any finding that might pose a risk to the participant.
* MRI brain findings of prior cerebellar stroke or clinical stroke within 12 months before screening.
* History of brain surgery regardless of purpose.
* Any contraindications to undergoing brain MRI.
* History of, or ongoing, malignant disease, (with the exception of basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 12 months prior to screening). Participants with cancers in remission for longer than 5 years may be included.
* History of epilepsy or the occurrence of seizures within 3 years prior to screening.
* Evidence of untreated/unstable thyroid disease.
* Poorly controlled diabetes mellitus.
* History of alcohol or substance abuse within the past year prior to screening.
* Use of off-label drugs for ataxia within 4 weeks prior to screening.
* Prior enrollment in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 5 half-lives or 3 months, whichever is longer, prior to the screening visit.
* Any antiplatelet [except for aspirin up to 100 milligrams per day (mg/day)] or anticoagulant medication that cannot be safely interrupted for an lumbar puncture (LP) procedure.
* Any contraindications to LP procedures.
* Participants who are pregnant or currently breastfeeding and those intending to become pregnant during the study.
* Prior enrollment in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 3 months prior to screening visit.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Day 1 to Day 267
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Screening to Day 267
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a-life threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85
Area Under the Concentration Versus Time Curve, from Time of Dosing (Time = 0) to Infinity (AUCinf) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85
Area Under the Concentration Versus Time Curve, from Time of Dosing (Time = 0) to Time of the Last Measurable Effect (AUClast) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85
Maximum Observed Concentration (Cmax) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85
Time to Reach Maximum Observed Concentration (Tmax) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85
Elimination Half-Life (t½) of BIIB132 | Pre-dose and at multiple timepoints post-dose on Day 1 up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (20):
- United States (10):
  - University of California - Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Florida, Center for Movement Disorders, Gainesville, Florida
  - Movement Disorder Center Florida, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia Univeristy Medical Center, New York, New York
  - Pennsylvania Neurological Institute, Philadelphia, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - University of Washington, Seattle, Washington
- Germany (3):
  - UniversitaetsklinikumTübingen Neurologische Universitätsklinik, Tübingen, Baden-Wurttemberg
  - Deutsches Zentrum fuer Neurodegenerative Erkrankungen (DZNE), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Essen Klinik für Neurologie, Essen, North Rhine-Westphalia
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Netherlands (2):
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Radboudumc, Nijmegen
- Portugal (2):
  - Centro Hospitalar de Lisboa Norte, Lisbon
  - Centro Hospitalar do Porto, Porto
- United Kingdom (2):
  - University College London Hospital (UCLH), London, Greater London
  - Churchill Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/